CLINICAL TRIAL: NCT06639334
Title: A Quick Pathway for Patients With High pRobability of dislocatEd Hemi- or Total Hip Arthroplasty to Minimize the Time From Hospital aDmission to redUCtion of the prosthEsis
Brief Title: The Q-REDUCE Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University Hospital of Southern Denmark (Unknown)
Responsible Party: Principal Investigator, Lars Lykke Hermansen, MD, PhD, University of Southern Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24/34681
Record Dates: First submitted 2024-07-29; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: THA; Dislocation, Hip; PROM
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Standard pathway for THA/HE reduction
  Interventions: Other: Standard pathway for THA/HE prosthesis reduction
- Fast-track treatment (Experimental): Fasttrack pathway for THA/HE reduction
  Interventions: Other: Fasttrack pathway for THA/HE prosthesis reduction

INTERVENTIONS:
Other: Fasttrack pathway for THA/HE prosthesis reduction — The purpose of this study is to design a fast-track pathway for patients referred to the University Hospital of Southern Denmark, Esbjerg, with high probability of having a dislocated hip prosthesis with the primary aim to reduce the time from arrival to reduction and the total hospitalization time.
  The intervention is changed logistic and work pathways at the hospital that should reduce time to reduction significantly. For detailed description we refer to the uploaded protocol.
  Arms: Fast-track treatment
Other: Standard pathway for THA/HE prosthesis reduction — Standard treatment for a dislocated THA/HA at our institution is education in general anesthesia at the operating theater. For detailed description we refer to the uploaded protocol.
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to design a fast-track pathway for patients referred to the University Hospital of Southern Denmark, Esbjerg, with high probability of having a dislocated hip prosthesis with the primary aim to reduce the time from arrival to reduction and the total hospitalization time. Secondary aims are to

* investigate whether quicker prosthesis reduction influences on hip function and quality of life afterwards
* reduce the pain experience immediately and in the long term
* increase patient satisfaction

without changing the overall complication rate and readmission/mortality

ELIGIBILITY:
Inclusion Criteria:

* a history of either a THA or a HA in combination with at least one of the following terms
* having sustained a sudden, incorrect movement or twist in the hip joint in either a bending, sitting or supine position leading to inability to stand or walk
* misalignment of the concerned lower extremity (typically shortened, with inward/outward rotation)

Exclusion Criteria:

* recurrent dislocations during the same hospital admission (already "in the house")
* anticipated difficult airway by the attending anesthesiologist
* anticipated need for extended respiratory or hemodynamic monitoring by the attending anesthesiologist
* American Society of Anesthesiologists (ASA) score > 3
* Body Mass Index (BMI) > 40
* active drug abuse
* contraindication for Propofol or Esketamine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Time from arrival at the emergency entrance to prosthesis reduction | 1 year

SECONDARY OUTCOMES:
Total hospitalization time from arrival to discharge | 1 year
Intra-operative complications (fracture, unsuccessful reduction, aspiration, need for mask ventilation and/or intubation, others) | 1 year
Post-operative complications (cardiac, pulmonal, thrombo-embolic events, nerve damage, re-dislocation, others) during hospitalization | 1 year
30 days re-admission | 30 days
30- and 90-days mortality | 30 and 90 days
Hip-related pain measured by a 10-digit numeric rating scale (NRS) | Day 0, 1, 3, 7, 14 and 30
  Evaluated from 1 (best) to 10 (worst).
Patient-reported outcome (PRO) using the Hip disability and Osteoarthritis Outcome Score (HOOS), | Day 0, 14, 90, 180 and 365
  Evaluated from 0 (worst) to 100 (best).
Health-related quality of life using the EQ-5D questionnaire | Day 0, 14, 90, 180 and 365
Patient satisfaction | During hospital admission, day 1.
  Consists of four self-developed questions.
Time consumption by the involved staff (orthopedic, anesthetic, radiology staff etc.) | 1 year
Total hospital costs during admission | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eggers Rasmussen L, Forberg Almas T, Kuhne-Qvist PJ, Beese Dalby R, Biesenbach P, Lykke Hermansen L. Quick pathway for patients with high pRobability of dislocatEd hemiarthroplasty or total hip arthroplasty to minimise the time from hospital aDmission to redUCtion of the prosthesis (Q-REDUCE): protocol for a prospective cohort study. BMJ Open. 2025 Jul 7;15(7):e091791. doi: 10.1136/bmjopen-2024-091791. PMID 40623887

DOCUMENTS (1):
  • Study Protocol (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT06639334/Prot_000.pdf